CLINICAL TRIAL: NCT06212336
Title: Efficacy, Tolerability and Safety of New or Repurposed Drugs Against Lassa Fever in West African Countries
Brief Title: ISTH/ANRS 0409s INTEGRATE Lassa Fever Study
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Irrua Specialist Teaching Hospital (Other)
Collaborators: Alliance for International Medical Action (Other); University of Bordeaux (Other); Bernhard Nocht Institute for Tropical Medicine (Other Government); Federal Medical Centre, Owo (Industry); Programme PAC-CI, Site ANRS-MIE de Côte d'Ivoire (Other); Fondation pour la Recherche Scientifique, Benin (Unknown); Médecins Sans Frontières, Belgium (Other); Alex Ekwueme Federal University Teaching Hospital (Other); Donka Hospital, Conakry (Unknown); Centre de Recherche Médicale de Lambaréné (Other); University of Hamburg-Eppendorf (Other); Phebe Hospital, Liberia (Unknown); University of North Carolina (Other); ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ISTH/ANRS 0409s INTEGRATE
Record Dates: First submitted 2023-09-22; First posted 2024-01-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Lassa Fever
Keywords: emerging infectious diseases; viral hemorrhagic fever; AFRICA; adult; adolescent
MeSH Terms: conditions — Lassa Fever; Communicable Diseases, Emerging; Hemorrhagic Fevers, Viral | interventions — favipiravir; Ribavirin; Standard of Care; Dexamethasone

STUDY DESIGN:
Intervention Model Description: a) Arms
  Intervention/ treatement
  Arm 1: SCD: ribavirin Arm:2 Favirpiravir 1600 Arm 3: Favipiravir 1200+ribavirin Arm 4: Ribavirin + dexamethasone Arm 5: ARN-75039 high dose (100) Arm 6: ARN-75039 low dose (50)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Favipiravir 1600 (Experimental): Oral favipiravir: 2400 mg BID D1; 1600 mg BID D2-D10
  Interventions: Drug: Favipiravir
- Ribavirin (Active Comparator): Intravenous ribavirin (Irrua regimen - 100 mg/kg Day 1 (dose is divided: 2/3 stat, 1/3 8 hours later, maximum dose is 7g/day) then 25 mg/kg single dose days 2-7, 12.5 mg/kg single dose days 8-10).
  Interventions: Drug: Favipiravir
- Favipiravir 1200 + ribavirin (Experimental): Oral favipiravir: 2400 mg BID D1; 1200 mg BID D2-D10 Intravenous ribavirin (Irrua regimen - 100 mg/kg Day 1 (dose is divided: 2/3 stat, 1/3 8 hours later, maximum dose is 7g/day) then 25 mg/kg single dose days 2-7, 12.5 mg/kg single dose days 8-10).
  Interventions: Drug: Favipiravir; Drug: Ribavirin
- Ribavirin + dexamethasone (Experimental): IV ribavirin, Irrua regimen IV or oral dexamethasone 6mg/day (For the first 48 hours, dexamethasone will be given intravenously (i. Afterwards, a switch to oral dexamethasone (same dosage) is permitted at the discretion of the study physician.)
  Interventions: Drug: Ribavirin; Drug: Dexamethasone
- ARN-75039 high dose (Experimental): • ARN-75039 high dose
  * D1: 300mg (morning), 200mg (evening)
  * D2: 200mg BID
  * D3-10: 100mg BID
  Interventions: Drug: ARN-75039 high dose
- ARN-75039 low dose (Experimental): • ARN-75039 low dose
  * D1: 150mg (morning), 100mg (evening)
  * D2: 100mg BID
  * D3-10: 50mg BID
  Interventions: Drug: ARN-75039 low dose

INTERVENTIONS:
Drug: Favipiravir — Interventional Medicinal Product (IMP)
  Arms: Favipiravir 1200 + ribavirin; Favipiravir 1600; Ribavirin
Drug: Ribavirin — Control arm
  Other Names: Standard of care
  Arms: Favipiravir 1200 + ribavirin; Ribavirin + dexamethasone
Drug: Dexamethasone — Interventional Medicinal Product (IMP)
  Arms: Ribavirin + dexamethasone
Drug: ARN-75039 high dose — Investigational Medicinal Product
  Arms: ARN-75039 high dose
Drug: ARN-75039 low dose — Investigational Medicinal Product
  Arms: ARN-75039 low dose

SUMMARY:
Lassa fever (LF) is a viral haemorrhagic fever responsible of 5000 deaths per year in West Africa, with in-hospital mortality at 12%. Transmission to humans occurs mainly via direct or indirect exposure to excreta from the rodent reservoir, mainly made up of Mastomys natalensis . Less frequently, LASV may also be transmitted from human to human and cause nosocomial outbreaks. Ribavirin is the only treatment available with worrying toxicity, questionable efficacy and low access because of its high cost. Consequently, there is an urgent need for new drugs to treat LF patients. The Research and Development (R&D) Blueprint of the World Health Organization (WHO) has included LF in the list of priority diseases for urgent research and development.

The INTEGRATE consortium is an unprecedented international collaboration on Lassa fever of 15 partners from 10 countries across West Africa, Europe and North America and across several disciplines (epidemiological researchers, social scientists, medical health facility professionals, humanitarian actors, etc.).

DETAILED DESCRIPTION:
The INTEGRATE study is a platform, multinational, multicentre, sequential, seamless phase II-III, controlled, randomised, superiority trial in open-label parallel arms. Three arms will be assessed and compared to the SCD. Its primary objective is to compare the efficacy of each Investigational Medical Product (IMP) to Standard of Care Drug (SCD) to prevent death or organ failure in hospitalized patients with confirmed LF. Secondary objectives will be i) to compare the safety and tolerability of each IMP and SCD, ii) to compare the efficacy of each IMP and SCD on clinical, virological and biological parameters, iii) to describe the pharmacokinetics of each IMP and iv) to develop a pharmacokinetics / pharmacodynamics model for each IMP informing about optimal dosing regimens and dose-response relationship.

1. Objectives

   1.1 Primary objective The primary objective of the trial is to compare the efficacy of each IMP and SCD to prevent death or organ failure in hospitalized participants with confirmed LF.

   1.2. Secondary objectives
   * To compare the safety and tolerability of each IMP and SCD
   * To compare the efficacy of each IMP and SCD on clinical, virological and biological parameters
   * To describe the pharmacokinetics of each IMP
   * To develop a pharmacokinetics / pharmacodynamics model for each IMP informing about optimal dosing regimens and dose-response relationship
2. Design

   * Phase II: comparative controlled design
   * Phase III: Whitehead's sequential double triangular design
3. Sample size:

   In the current version of the protocol (if all sub-protocols start at once):
   * 3 IMPs go into phase III: N= 732
   * 2 IMPs go into phase III: N= 585
   * 1 IMP go into phase III: N= 438
4. Duration

   * Hospitalization: 10 days
   * Follow-up: 28 days

ELIGIBILITY:
1. General

   Inclusion criteria
   * Clinical disease with signs and symptoms suggestive for LF
   * Positive plasma LASV RT-PCR
   * Participant requires hospitalization per the local guidelines
   * Participant or their legally authorized representative is able and willing to sign the informed consent

   Exclusion criteria
   * Unwilling to provide informed consent
   * Positive pregnancy test
   * Unwilling to provide informed consent
   * History of allergic reaction or other contra-indication to ribavirin according to the Reference safety document
   * Received drug therapy for Lassa fever (excluding supportive care) prior to inclusion
   * Has received a vaccine against LF
2. Sub-protocols

   2.1 Favipiravir high dose sub-protocol

   Inclusion criteria • Age ≥ 18 years old

   Exclusion criteria • Pregnancy (evidenced by positive urine pregnancy test in women of child-bearing potential)
   * Treatment contraindicated with favipiravir according to the Reference safety document
   * Pre-existing liver failure
   * Severe symptomatic gout/hyperuricemia
   * History of QT prolongation or arrhythmia or other cardiac disorders
   * PR interval ≥ 200 ms
   * Hypersensitivity to excipients
   * Inability to take oral drug (e.g. encephalopathy, severe vomiting)

   2.2. Favipiravir-Ribavirin sub-protocol

   Inclusion criteria

   • Age ≥ 18 years old

   Exclusion criteria
   * Pregnancy (evidenced by positive urine pregnancy test in women of child-bearing potential)
   * Treatment contraindicated with favipiravir according to the Reference safety document
   * Pre-existing liver failure
   * Severe symptomatic gout/hyperuricemia
   * History of QT prolongation or arrhythmia or other cardiac disorders
   * PR interval ≥ 200 ms
   * Hypersensitivity to excipients
   * Inability to take oral drug (e.g. encephalopathy, severe vomiting)

   2.3. Dexamethasone sub-protocol

   Inclusion criteria • Age ≥ 12 years old

   Exclusion criteria

   • Pregnancy (evidenced by positive urine pregnancy test in women of child-bearing potential)

   • Known intolerance and contra-indications to ribavirin or dexamethasone

   • Patients who already received a corticosteroid within the preceding 7 days

   2.4 ARN-75039 subprotocols

   Exclusion criteria • History of severe gastrointestinal disease

   • History of chronic generalized pruritus
   * History of severe chronic liver disease
   * History of severe cardiac disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1755 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Death | Day 28
  Proportion of participants death definition by Y/N measure
  Clinical aggravation is defined as the first occurrence of one of the following conditions, at any time point between baseline and Day 14 (included):
  Death, or
  Increase (+1 or +2) in the number (0, 1 or 2) of organ failures among:
  Renal failure: KDIGO stage 3 Respiratory failure: SpO2/FiO2* ≤ 315 Cardiovascular failure: MBP** < 65 mmHg or SBP < 90 mmHg (measured twice with a time interval of 10 min) and lactate > 2 mmol/L Analysis per component Proportion of participants with a newly occurring component of the composite primary endpoint between Day 0 and Day 14.
  Sensitivity analyses Proportion of participants presenting no clinical aggravation between baseline and Day 14, with varying thresholds on the definitions of organ failures or adding different organ failures definition (e.g. neurologic, hepatic, hematologic, etc.).
New onset of acute kidney failure | Between Day 0 and Day 10
  Proportion of participants a new onset of acute kidney failure . Definition by KDIGO 3 measure. 3.0 times baseline, OR increase in serum creatinine to ≥4.0 mg/dl (≥353.6 mmol/l).
  The composite endpoint assesses the new onset of an event from D0
New onset of acute respiratory failure | Between Day 0 and Day 10
  Proportion of participants a new onset of acute respiratory failure. Definition by SpO2/FiO2 ≤ 315 measure The composite endpoint assesses the new onset of an event from D0
New onset of shock | Between Day 0 and Day 10
  Proportion of participants a New onset of shock. Mean Blood Pressure (MBP) < 65 mmHg or Systolic Blood Pressure (SBP) < 90 mmHg (measured twice with a time interval of 10 min) and lactate > 2 mmol/L measured at the same time The composite endpoint assesses the new onset of an event from D0

SECONDARY OUTCOMES:
Safety of each IMP and SCD | Between Day 0 and Day 10
  Proportion (events and participants with at least one event) of:
  * Adverse Event* grade 3 and higher
  * Serious Adverse Event
  * Adverse Event of Special Interest
Safety of each IMP and SCD | Day 0, Day 28
  Proportion (events and participants with at least one event) of:
  Adverse Event* grade 3 and higher
  * Serious Adverse Event
  * Adverse Event of Special Interest
Organ failure from composite primary endpoint | Between Day 0 and Day 10
  Proportion of participants with a newly occurring component of the composite primary endpoint
New onset of Acute Kidney Injury | Between Day 0 and discharge
  Proportion of participants meeting KDIGO ≥ 2 or initiation of renal replacement therapy parameters
New onset of CVPU or seizure | Between Day 0 and Discharge
  Proportion of participants with CVPU or seizure
New onset of Bleeding | Between Day 0 and Discharge
  Proportion of participants meeting WHO bleeding scale grade 2 or above
New onset of Severe anaemia | Between Day 0 and Discharge
  Proportion of participants with Hb level < 8 g/dL
New onset of liver failure | Between Day 0 and Discharge
  Proportion of participants with AST or ALT ≥ 3 ULN
New onset of clinical severity score | Between Day 0 and Discharge
  Proportion of participants with a NEWS2 score ≥7
Intensive care strategies - oxygen therapy | Between Day 0 and Discharge
  Proportion of participants having received oxygen therapy
Intensive care strategies - RRT | Between Day 0 and Discharge
  Proportion of participants having received RRT
Intensive care strategies - blood transfusion | Between Day 0 and Discharge
  Proportion of participants having received blood transfusion
Intensive care strategies- inotropes or vasopressors | Between Day 0 and Discharge
  Proportion of participants having received inotropes or vasopressors
the viral clearance - Change in LF RT-PCR Ct | Day 3, Day 5, Day 7, Day 9
  value (for each target gene) from D0
the viral clearance - Change in LASV viral | D01-D10
  titer from D0
viral clearance - LASV RT-PCR | D01- D10
  <LLQ
Pharmacokinetics (phase II only) | Between Day 0 and Day 10
  • Peak concentration (Cmax)
Pharmacokinetics (phase II only) | Between Day 0 and Day 10
  • Time to peak concentration (Tmax)
Pharmacokinetics (phase II only) | Between Day 0 and Day 10
  • Area under the curve
Pharmacokinetics (phase II only) | Between Day 0 and Day 10
  • Half-life
Pharmacokinetics (phase II only) | Between Day 0 and Day 10
  • Clearance
Pharmacokinetics (phase II only) | Between Day 0 and Day 10
  • Volume(s) of distribution
PK/PD (phase II only) | Between Day 0 and Day 10
  • Prediction of initial viral load and slope of decline
PK/PD (phase II only) | Between Day 0 and Day 10
  • Optimal dosing regimen with PK/PD modelling
LASV RT-PCR | D28 if participants have a positive RT PCR at discharge
  LASV RT-PCR (Ct value)
Peak CRP (Phase II stage only) | D01-D10
  Peak CRP level (mg/L)
Time to first LASV RT-PCR <LLOQ | D01-D10
  Time to first LASV RT-PCR <LLOQ (days)

OTHER OUTCOMES:
Viral resistance parameters | Between Day 0 and Day 10
  Frequency of LASV resistance mutations

CONTACTS AND LOCATIONS:
Overall Officials: Marie MD JASPARD, MD, Study Director — ALIMA - The Alliance for International Medical Action - Paris, France; Sylvanus OKOGBENIN, MD, Principal Investigator — Irrua Specialist Teaching Hospital Irrua - Edo State, Nigeria; Michael RAMHARTER, MD, Study Chair — Bernhard Nocht Institute for Tropical Medicine Bernhard-Nocht-Hamburg, Germany
Locations (4):
- Phebe Hospital, Suacoco, Bong County, Liberia
- Nigeria (3):
  - Irrua Specialist Teaching Hospital, Irrua, Edo
  - Federal Medical Center Owo, Owo, Ondo State
  - Abubakar Tafawa Balewa University Teaching Hospital, Bauchi

IPD SHARING:
Plan to Share IPD: Undecided